CLINICAL TRIAL: NCT06885242
Title: Efficacy and Safety of Cyclopentolate Microdrops for Cycloplegic Refraction in Children: a Non-inferiority Crossover Randomized Controlled Trial
Brief Title: Efficacy and Safety of Cyclopentolate Microdrops for Cycloplegic Refraction in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Nanodropper, Inc. (Industry)
Responsible Party: Principal Investigator, Asimina Mataftsi, Professor in Ophthalmology, Paediatric Ophthalmology and Strabismus, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 383/19-06-2024
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Cycloplegic Refraction
Keywords: microdrops; cycloplegia; refraction; cyclopentolate; children

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study Group (Experimental): Cycloplegia with microdrops
  Interventions: Device: Microdrop instillation of cyclopentolate 1%
- Control Group (Active Comparator): Cycloplegia with standard drops
  Interventions: Device: Standard drop instillation of cyclopentolate 1%

INTERVENTIONS:
Device: Microdrop instillation of cyclopentolate 1% — 1 drop administered through the Nanodropper device adapted to the commercially available multi-dose dropper bottle
  Arms: Study Group
Device: Standard drop instillation of cyclopentolate 1% — 1 drop administered directly through the commercially available multi-dose dropper bottle
  Arms: Control Group

SUMMARY:
The purpose is to test the hypothesis that microdrop instillation of cyclopentolate 1% is non-inferior to standard of care, i.e., standard drop instillation of cyclopentolate 1%. Comparison, also, will be made to the subsequent adverse events.

DETAILED DESCRIPTION:
A non-inferiority, crossover, randomized controlled trial will be conducted for this purpose. Participants will be randomly assigned to receive either a) microdrops on their first and standard drops on their second screening examination a week later (M/S group), or b) standard drops first and microdrops a week later (S/M group). Microdrops will be instilled using the Nanodropper® device, while standard drops will be instilled directly through the commercially available plastic multidose mydriatic dropper bottle. For all participants, the eyedrop will be firstly instilled in the right eye and this will be the eye that will be used for the analyses. Written informed consent will be obtained from the parents/guardians for the children's enrollment.

ELIGIBILITY:
Inclusion Criteria:

Children aged 4-16 years old, who require cycloplegic refraction measurements in the context of regular ophthalmological examination as outpatients in the 2nd Department of Ophthalmology of AUTh at a tertiary center in Northern Greece.

Exclusion Criteria:

1. Inability for the child to cooperate with autorefractometer
2. Difficulties for the family to attend the follow-up visit
3. Known allergic reaction to cyclopentolate or to any of the other ingredients of this solution
4. Presence of any contraindication for the child to receive cyclopentolate eyedrops (e.g. neurological disease of concern)

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Cycloplegic refraction: diopters of spherical equivalent | 40 minutes post-instillation
  The difference in spherical equivalent (SE) after microdrop and standard drop instillation (cycloplegic efficacy)

SECONDARY OUTCOMES:
Heart rate: bpm | 40 minutes post-instillation
  The difference in heart rate after microdrop and standard drop instillation (safety outcome)
Flushing: absent, minor, major | 40 minutes post-instillation
  The difference in the number of patients who experience flushing after microdrop and after standard drop instillation (safety outcome)
Behavioral changes: yes or no | 40 minutes post-instillation
  The difference in the number of patients who experience behavioral changes after microdrop and after standard drop instillation (safety outcome)
Sleepiness: yes or no | 40 minutes post-instillation
  The difference in the number of patients who experience sleepiness after microdrop and standard drop instillation (safety outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Seliniotaki AK, Tziola T, Lithoxopoulou M, Tzamalis A, Ziakas N, Mataftsi A. Optimizing instilled drug delivery: a scoping review of microdrops in ophthalmology. Graefes Arch Clin Exp Ophthalmol. 2025 Jul;263(7):1765-1787. doi: 10.1007/s00417-025-06773-1. Epub 2025 Feb 26. PMID 40011238
- [Background] Hoppe CB, Yonamine S, Kao BW, Turner ML, Ou Y, Han Y, Keenan JD, Oatts JT. Randomized Trial to Evaluate the Efficacy of the Nanodropper Device for Pupillary Dilation and Cycloplegia in Children. Ophthalmology. 2023 Mar;130(3):324-330. doi: 10.1016/j.ophtha.2022.10.016. Epub 2022 Oct 22. PMID 36280185
- [Background] Noske W. Cycloplegic refraction using atropine minidrops. Strabismus. 1993;1(1):17-23. doi: 10.3109/09273979309033849. PMID 21314515